CLINICAL TRIAL: NCT02106637
Title: Early In-hospital Initiation of Pharmacotherapy for Smoking Cessation, Concomitant With Nurse-Led Support, in Patients After an Acute Coronary Syndrome (ACS)
Brief Title: Early In-hospital Initiation of Pharmacotherapy for Smoking Cessation, Patients After ACS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Hadassah Medical Organization (Other); Barzilai Medical Center (Other)
Responsible Party: Principal Investigator, Prof. Ilan Goldenberg, MD, Prof. Ilan Goldenberg, MD, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHAMPIX (CHANTIX)
Record Dates: First submitted 2014-03-27; First posted 2014-04-08 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Acute Coronary Syndrome; Smoking Cessation
Keywords: ACS; Cessation
MeSH Terms: conditions — Acute Coronary Syndrome; Smoking Cessation | interventions — Varenicline; Time

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- study groups (Active Comparator): study groups will receive Varenicline
  Interventions: Drug: Varenicline
- control group (Placebo Comparator): Participants allocated to the control group will receive placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Varenicline — drug will be initiated during hospitalization and continued for 12 weeks following discharge
  Other Names: CHAMPIX; CHANTIX
  Arms: study groups
Drug: placebo — placebo
  Other Names: Matching placebo for 12 weeks duration
  Arms: control group

SUMMARY:
The hypothesis of this study is that combination of Varenicline treatment with nurse-led hospital support during hospitalization and after discharge will result in clinically significant higher long term abstinence rates in smokers with ACS, as compared with nurse led support and placebo, without a significant increase in the risk of adverse events.

DETAILED DESCRIPTION:
Smokers hospitalized with Acute Coronary Syndrome (ACS) are at high risk for ischemic events or death. Over two thirds of patients continue to smoke after acute myocardial infarction.

Study objectives will evaluate safety and efficacy of Varenicline vs. placebo in hospitalized ACS patients complemented by nurse-led support. Interventions will continue following discharge for the duration of 12 weeks.

The primary efficacy outcome measure is continuous abstinence rate at 1 year after hospitalization as assessed by self-reporting and verified by CO breath test.

The proposed study is a prospective, double blind, randomized, placebo controlled, multi-center study. Overall 300 patients will be recruited, randomly allocated to active and placebo treatment groups that will receive nurse-led support by trained staff.

Hospitalized ACS smokers will be evaluated by the protocol inclusion/exclusion criteria. Patient's demographics, medical and laboratory data will be obtained including Fagestrom tobacco addiction questionnaire and digitally captured. Participants will be randomly allocated to study groups and will receive, Varenicline or placebo, which will be initiated on the last day of hospitalization and continued for 12 weeks after discharge. Additionally, a structured nurse-led behavioral support program for smoking cessation will be initiated during hospitalization, followed by telephone calls that will provide motivational support and an interview exploring protocol adherence, side effects, changes in health status and smoking status.

All patients will be re-assessed at one, 3 and 12 -months post discharge. Follow-up visits will comprise of a physical examination, adverse event assessment and CO breath testing.

Cardiovascular diseases are the leading cause of death in Western countries, and cigarette smoking has a clear cause-and -effect relationship with atherosclerotic disease (1). Smokers hospitalized with Acute Coronary Syndrome (ACS) are at high risk for subsequent ischemic events and present 50% higher chance of death in the first 2 years (2). Nevertheless, over two thirds of patients continue to smoke after an acute myocardial infarction. Varenicline has been shown to be highly effective smoking cessation intervention (4), yet concerns have been raised regarding safety in coronary patients (5).

A significant number of eligible patients do not receive structured smoking cessation interventions following ACS. Initiation of secondary prevention interventions during hospital stay has been shown to be highly effective for other key secondary prevention interventions (i.e. statins, beta blockers).

Moreover, combination of Varenicline treatment with nurse-led hospital support, initiated early during hospitalization is expected to result in better adherence and better long-term abstinence rates in smokers with a recent ACS.

This proposed study would be the first Israeli trial with Varenicline.

ELIGIBILITY:
Inclusion Criteria:

* Stable clinical condition following a recent (< 10 days) ACS event
* Active smoking status 30-days prior to ACS
* Age > 21
* Life expectancy >1 year

Exclusion Criteria:

I. Severe pulmonary disease (FEV1 < 30% predicted ) II. End stage renal failure (eGFR < 20 ml/min/m2) III. Uncontrolled depression or history of psychosis or bipolar disorder or active substance abuse IV. Uncontrolled stage IV hypertension V. Un-resolved life threatening arrhythmia VI. Planned surgical intervention (within < 3 months) VII. Known hypersensitivity to study drug components VIII. Inability to comply with study protocol IX. Active malignancy other than basal cell carcinoma (BCC) X. End-stage congestive heart failure - NYHA IV or decompensated heart failure XI. Pregnancy or lactation

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy and Safety endpoint: | within 12 month from enrollment
  Continuous abstinence rate (CAR) from smoking 1-year after hospitalization as determined by self-reporting and verified by CO testing. Only the combination of the two will be considered as achieving CAR .
  Non inferior serious adverse event (SAE) rate, defined as: event rate in the intervention group compared to the placebo (SAE according to the FDA definitions) group at 12 months. An interim analysis will be preformed after 33% and 66% of patients have been finished the follow-up duration.

SECONDARY OUTCOMES:
Secondary Outcomes - Weight change | Within 12 month from enrollmen
  Weight change in the intervention group vs. placebo , Baseline vs. 12 month visit
Smoking abstinence at 1 and 6 months | 1 and 6 months after randomization
  CAR at 1- and 6-month visits as reported and verified by CO breath analysis

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Goldenberg, Prof., Study Director — Sheba Medical Center; Haim Lotan, MD, Principal Investigator — Hadassa medical organisation; Haim Yosefi, MD, Principal Investigator — Barzili Medical Center; Robert Klempfner, MD, Study Director — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Derived] Streck JM, Rigotti NA, Livingstone-Banks J, Tindle HA, Clair C, Munafo MR, Sterling-Maisel C, Hartmann-Boyce J. Interventions for smoking cessation in hospitalised patients. Cochrane Database Syst Rev. 2024 May 21;5(5):CD001837. doi: 10.1002/14651858.CD001837.pub4. PMID 38770804
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273